CLINICAL TRIAL: NCT07216157
Title: The NoSeal Trial - Nasal Outcome Study Evaluating Artificial Leak-Sealing: A Prospective, Randomized, Controlled, Single-Blinded, Single-Center Clinical Trial Comparing Fibrin Glue (Tisseel®) and a Two-Component Synthetic Polymer Sealant (PEI/PEG, Adherus®) Versus No Sealant for the Prevention of Cerebrospinal Fluid Leak and Promotion of Wound Healing Following Endonasal Skull Base Surgery, Designed in Accordance With the SPIRIT 2025 Guidelines
Brief Title: NoSeal Trial: Comparing Sealants Versus No Sealant for Preventing CSF Leak After Endonasal Skull Base Surgery
Acronym: NoSeal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Principal Investigator, Wojciech Czyżewski, Wojciech Czyżewski MD, PhD, Neurosurgery Specialist, Principal Investigator, Maria Sklodowska-Curie National Research Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIO-NS2025
Record Dates: First submitted 2025-09-28; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-07

CONDITIONS: CerebroSpinal Fluid (CSF) Leak
Keywords: csf; pituitary adenoma; csf leak; sealant
MeSH Terms: conditions — Pituitary Neoplasms; Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- No Sealant - Standard Multilayer Closure (Experimental): Patients in this arm will receive standard multilayer closure without the use of any sealant. Closure will involve mucosal flap repositioning and hemostatic agents (e.g., Surgicel®, TachoSil®), in accordance with standard endoscopic skull base reconstruction techniques.
  Interventions: Procedure: Standard multilayer closure without sealant
- Fibrin Glue - Tisseel® Application (Experimental): Patients will undergo standard multilayer closure followed by application of fibrin sealant (Tisseel®). This arm evaluates the effect of biologic tissue glue in preventing postoperative CSF leaks and promoting wound healing following endonasal skull base surgery.
  Interventions: Device: Fibrin sealant application
- Synthetic Sealant - Adherus® Application (Experimental): This arm involves standard multilayer closure followed by the application of a two-component synthetic polyethylene glycol-based sealant (Adherus®). The objective is to evaluate the synthetic agent's efficacy and cost-effectiveness in reducing postoperative CSF leaks.
  Interventions: Device: Synthetic polyethylene glycol-based sealant

INTERVENTIONS:
Procedure: Standard multilayer closure without sealant — Patients will undergo standard skull base reconstruction using mucosal flap repositioning and absorbable hemostatics (e.g., Surgicel®, TachoSil®), without application of any fibrin or synthetic sealant. This serves as the control group for comparison with sealant-assisted closures.
  Other Names: No-sealant technique; Control arm
  Arms: No Sealant - Standard Multilayer Closure
Device: Fibrin sealant application — Following standard multilayer closure, patients in this group will receive topical application of a fibrin-based biological sealant (Tisseel®). The intervention aims to assess its effectiveness in preventing postoperative cerebrospinal fluid (CSF) leak and promoting mucosal healing after endoscopic endonasal skull base surgery.
  Other Names: Tisseel®; Fibrin glue; Human fibrinogen/thrombin sealant
  Arms: Fibrin Glue - Tisseel® Application
Device: Synthetic polyethylene glycol-based sealant — After standard multilayer closure, a synthetic two-component sealant (Adherus®, composed of polyethylene glycol and polyethylenimine) will be applied to reinforce the reconstruction site. This group is used to evaluate the efficacy and safety of synthetic sealant in preventing CSF leaks and supporting wound healing.
  Other Names: Adherus®; PEI/PEG sealant; Synthetic dural sealant
  Arms: Synthetic Sealant - Adherus® Application

SUMMARY:
Postoperative cerebrospinal fluid (CSF) leak is a significant complication of endoscopic endonasal approaches (EEA) to the skull base. The use of tissue sealants such as fibrin glue (Tisseel) or synthetic agents (PEI/PEG) is widespread in surgical practice, however, recent high-quality evidence challenges their clinical benefit and cost-effectiveness. This study aims to investigate whether the routine use of sealants in patient with peri-operatively assessed low CSF leak risk, significantly improves outcomes over no sealant use, to guide more cost- effective, evidence-based closure strategies. To the best of our knowledge, the present study is the first randomized clinical trial to evaluate the necessity and comparative effectiveness of fibrin and synthetic sealants versus no sealant in preventing postoperative CSF leaks following endoscopic endonasal surgery in low-post operative CSF leak risk patients.

DETAILED DESCRIPTION:
Introduction Postoperative cerebrospinal fluid (CSF) leak is a significant complication of endoscopic endonasal approaches (EEA) to the skull base. The use of tissue sealants such as fibrin glue (Tisseel) or synthetic agents (PEI/PEG) is widespread in surgical practice, however, recent high-quality evidence challenges their clinical benefit and cost-effectiveness. This study aims to investigate whether the routine use of sealants in patient with peri-operatively assessed low CSF leak risk, significantly improves outcomes over no sealant use, to guide more cost- effective, evidence-based closure strategies. To the best of our knowledge, the present study is the first randomized clinical trial to evaluate the necessity and comparative effectiveness of fibrin and synthetic sealants versus no sealant in preventing postoperative CSF leaks following endoscopic endonasal surgery in low-post operative CSF leak risk patients. Materials and Methods This is a prospective, randomized, controlled, single-center clinical trial conducted at the Maria Skłodowska-Curie National Research Institute of Oncology in Warsaw, Poland.

Adult patients scheduled for endoscopic endonasal surgery (EES) will first undergo screening based on medical history and detailed radiological evaluation. Those who meet all predefined inclusion and exclusion criteria will be enrolled and randomized preoperatively using a computer-generated allocation sequence into one of three treatment arms: (1) no sealant (standard multilayer closure), (2) fibrin glue application (Tisseel®), or (3) synthetic polyethylene glycol-based sealant (Adherus®). Following randomization, surgery will be performed in accordance with the assigned intervention. The primary endpoint is the incidence of postoperative cerebrospinal fluid (CSF) leak within 3 months. Secondary outcomes include endoscopic evaluation of mucosal healing at 6 weeks and 3 months, postoperative complication rates (e.g., meningitis, pneumocephalus), reoperation rate, patient-reported quality of life, and a cost-effectiveness analysis comparing sealant use to standard closure. The study is designed and will be reported in accordance with the SPIRIT 2025 (Standard Protocol Items: Recommendations for Interventional Trials) guidelines to ensure methodological transparency and reproducibility. Results Initial enrollment includes a target of 225 patients (75 per arm). Interim data analysis focuses on early healing parameters, safety profiles, and cost metrics. Hypothesis testing will determine if either sealant significantly reduces CSF leak rates compared to no sealant and whether the marginal benefit justifies routine use in all patients. Exploratory endpoints include biomaterial handling characteristics and surgeon-reported usability. Conclusion The NoSeal Trial addresses a critical gap in evidence regarding the necessity and comparative performance of sealants in skull base reconstruction. By evaluating both clinical outcomes and economic impact, the study seeks to optimize surgical protocols and improve the safety and efficiency of endonasal neurosurgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for endoscopic endonasal surgery involving standard skull base reconstruction
* Informed written consent obtained prior to enrollment
* Hemodynamic and electrolyte stability before surgery
* Procedure expected to be completed without use of high-flow intraoperative CSF diversion techniques

Exclusion Criteria:

* Revision surgery or extended endoscopic approaches requiring complex reconstruction (e.g., clival or cribriform defects)
* Tumors requiring complex sella reconstruction from the start
* Preoperative hydrocephalus
* Known allergy to fibrin-based or synthetic sealant components
* Active sinus infection or systemic inflammatory disease
* Prior radiotherapy to the sellar or parasellar region
* Uncontrolled diabetes mellitus (HbA1c > 7.0%)
* Participation in another interventional trial that may influence wound healing or CSF assessment
* Radiologic signs of chronic intracranial hypertension or hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative cerebrospinal fluid (CSF) leak within 90 days | 90 days
  Postoperative CSF leak will be assessed clinically and endoscopically at multiple time points (Day 2, Day 30, Day 90). A leak will be defined as visible or symptomatic leakage of cerebrospinal fluid from the nasal cavity, confirmed by clinical exam and/or imaging when necessary. Assessment will be blinded and recorded using standardized diagnostic criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) to be shared will include:
  Demographics (age, sex) Preoperative imaging risk features Intraoperative findings (CSF leak grade, reconstruction technique) Treatment allocation (sealant type or no sealant) Primary and secondary outcomes (e.g., CSF leak occurrence, mucosal healing scores, complication rates, SNOT-22 and VAS scores) Follow-up data at 4 and 12 weeks Reoperation status Adverse events
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified individual participant data (IPD) and supporting documentation will be available beginning 6 months after publication of the primary results and will remain accessible for up to 36 months.
Access Criteria: Access will be granted to qualified researchers affiliated with academic or non-commercial institutions who submit a methodologically sound research proposal. Access will include de-identified IPD and supporting documents (protocol, SAP, ICF, CSR, analytic code). Requests should be sent to the corresponding author. Data will be shared via secure institutional data-sharing platforms upon approval of the proposal and execution of a data use agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-23): https://cdn.clinicaltrials.gov/large-docs/57/NCT07216157/Prot_SAP_000.pdf